CLINICAL TRIAL: NCT00671151
Title: Molecular Mechanisms of COPD Exacerbations. Effect of Low-Dose Theophylline
Brief Title: Effects of Low-Dose Theophylline During Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Son Dureta (Other)
Collaborators: Fondo de Investigación Sanitaria (FIS) (Unknown); Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Borja G Cosio MD, Specialist in Respiratory Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: FIS042146
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2008-04

CONDITIONS: COPD
Keywords: COPD exacerbation; histone; steroid resistance; inflammation; theophylline
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Theophylline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Low-dose theophylline on top of standard therapy for COPD exacerbation
  Interventions: Drug: Theophylline
- 2 (No Intervention): Standard therapy for COPD exacerbation

INTERVENTIONS:
Drug: Theophylline — Theophylline 100 mg bid for 3 months
  Arms: 1

SUMMARY:
Molecular mechanisms of COPD exacerbations and the modulating effect of low dose theophylline on that inflammation are elucidated in this project. NF-kappa B-dependent pathway and acetylation status of nuclear histones are to be studied.Design: controlled, prospective and randomized study with or without theophylline, a potent HDAC activator.Objectives: 1) To determine NF-kB activation, histone deacetylase (HDAC) and histone acetyl-transferase (HAT) activity in sputum macrophages and blood monocytes during an episode of exacerbation and 3 months later, once stability is achieved. To correlate these measurements with inflammatory and oxidative stress markers and with pulmonary function and clinical variables. 2) To assess the effect of theophylline on previous molecular, functional and clinical data. Method: 25 patients with COPD will be recruited during an episode of exacerbation requiring hospitalization. NF-kB activation, HDAC and HAT activity, markers of inflammation and oxidative stress will be determined with specific assays. These determinations will be repeated once the patient is stable and compared with smokers and non smoker controls with normal lung function

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD according to GOLD guidelines
* Age between 40 and 75
* Admission to hospital due to COPD exacerbation

Exclusion Criteria:

* History of asthma
* Pulmonary embolism
* Pneumonia
* Other chronic inflammatory disease
* Patient on theophylline at the time of admission
* Patient on oral steroids at the time of admission

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
HDAC activity in alveolar macrophages | 3 months

SECONDARY OUTCOMES:
Lung function | 3 months
Inflammatory cytokine release in sputum and serum | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Borja G Cosio, MD, Principal Investigator — Hospital Universitario Son Dureta
Locations (1):
- Hospital Universitario Son Dureta, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Cosio BG, Tsaprouni L, Ito K, Jazrawi E, Adcock IM, Barnes PJ. Theophylline restores histone deacetylase activity and steroid responses in COPD macrophages. J Exp Med. 2004 Sep 6;200(5):689-95. doi: 10.1084/jem.20040416. Epub 2004 Aug 30. PMID 15337792
- [Derived] Cosio BG, Iglesias A, Rios A, Noguera A, Sala E, Ito K, Barnes PJ, Agusti A. Low-dose theophylline enhances the anti-inflammatory effects of steroids during exacerbations of COPD. Thorax. 2009 May;64(5):424-9. doi: 10.1136/thx.2008.103432. Epub 2009 Jan 21. PMID 19158122